CLINICAL TRIAL: NCT07157709
Title: Implementation of the Pain Management Toolkit in a Nursing Home
Brief Title: Implementation of the Pain Management Toolkit
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Medizinische Universität Graz, Institut für Pflegewissenschaft (Other)
Responsible Party: Principal Investigator, Manuela Hoedl, Univ.-Ass. Priv.-Doz. Dr.rer.cur. BSc MSc, Medizinische Universität Graz, Institut für Pflegewissenschaft
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EK Nr:1371/2024; CM-300 (Other Grant/Funding Number: Austrian Science Fund)
Record Dates: First submitted 2025-08-18; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Pain
Keywords: pain; pain management; implementation; toolkit; non-pharmacological; long term care
MeSH Terms: conditions — Pain; Agnosia | interventions — Exercise; Relaxation Therapy; Hypnosis; Patient Positioning; Osteogenesis, Distraction; Laughter Therapy; Massage; Music Therapy; Oils, Volatile

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- non-pharmcological interverntions to reduce pain (Experimental): non-pharmacological interventions will be administered in order to treat pain
  Interventions: Other: non-pharmacological interventions

INTERVENTIONS:
Other: non-pharmacological interventions — Care staff collaborate with residents to select the most suitable non-pharmacological intervention from the designated toolkit to reduce pain. It is imperative to pay attention to the resident's preferences and to ascertain which intervention they would like to attempt.
  Other Names: Empathic attention and communication; Physical exercise; Relaxation techniques; Self-hypnosis and fantasy journeys; Relieving pressure on affected body parts/positioning; Distraction; Promoting sleep; Psychological support; Cold application; Heat application; Wraps and compresses; Laughter therapy; Massage; Music; Aromatherapy: massage with essential oils; Aromatherapy: gargling with essential oils; Aromatherapy: inhalation of essential oils; Aromatherapy: lymphatic drainage with essential oils; Mindfulness exercises

SUMMARY:
The overall aim of this research study is to implement and evaluate the toolkitinto the nursing home by using scientific methods, which is cut down in specific aims.

1. To assess the effectiveness of the toolbox on

   1. staff outcomes
   2. pain management practice
   3. resident's outcomes
2. To identify potential barriers and facilitators of the implementation from the perspective of the staff
3. To investigate different outcomes of the implementation strategies

ELIGIBILITY:
Inclusion Criteria:

* presence of pain
* living in the collaborating nursing home

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Nursing staff self-efficacy in pain management (self-efficacy in pain management scale) | 1 year
  The self-efficacy from the nursing staff with regard to pain management will be assessed by the self-efficacy in pain management scale developed by Brunkert et al. in 2019.
Pain management process indicator: number of non-pharmacological measures | 1 year
  This data will be collected from the nursing home resident's record - the last 7 days will be assessed.
Pain management process indicator: number/dosage of pain medication | 1 year
  This data will be collected from the nursing home resident's record - the last 7 days will be assessed.
Resident's outcome indicator: frequency of pain | 1 year
  The frecquency of documented pain in the last 7 days will be assessed, by going through the nursing home resident's records.
Resident's outcome indicators: pain intensity | 1 year
  Pain intensity will be assessed by the documented pain in the nursing home resident's records. The most recent pain intensity score will be used.
Resident's outcome indicators: pain impairment (PEG scale) | 1 year
  The pain impairment will be assessed by using the PEG scale developed by Wander et al. in 2022.
Resident's outcome indicators: quality of life (VAS scale) | 1 year
  The EQ-5D VAS is an internationally well-known, valid and reliable instrument to assess quality of life in adults in will be used to assess health related quality of life.

SECONDARY OUTCOMES:
Staff's perception about implementation barriers (pCAT) | 1 year
  To assess staff's perception about implementaiton barrieres, the pCAT questionnaire will be used.
Staff's perception about implementation facilitators (pCAT) | 1 year
  To assess staff's perception about implemenation facilitators, the pCAT questionnaire will be used.

OTHER OUTCOMES:
Staff's perception about the appropriateness of the toolkit (IAM scale) | 1 year
  The Intervention Appropriateness Measure (IAM) scale will be used.
Staff's perception about the feasibility of the toolkit (IAM scale) | 1 year
  The Intervention Appropriateness Measure (IAM) scale will be used to assess staff's perception about the feasibility of the toolkit.
Penetration of the toolkit (FIM scale) | 1 year
  The Feasibility of intervention measure (FIM) scale will be used to assess the penetration of the toolkit.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No